CLINICAL TRIAL: NCT00447239
Title: The Effect of Intensive Insulin Therapy on the Incidence of Ventilator-Associated Pneumonia in Surgical Critically Ill Patients
Brief Title: The Effect of Intensive Insulin Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: gluco study
Expanded Access: Available
Record Dates: First submitted 2007-03-13; First posted 2007-03-14 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2007-03

CONDITIONS: the Maintenance of Normoglycemia; the Incidence of Ventilator Associated Pneumonia (VAP); Treatment Period in the Intensive Care Unit
Keywords: mechanical ventilated; surgical patients; pneumonia; blood glucose; insulin infusion; hospital stay
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: glucontrol (insulin therapy)

SUMMARY:
Aim. To determine whether the maintenance of normoglycemia decreases the incidence of ventilator associated pneumonia (VAP), reduces its treatment period and the length of stay in the intensive care unit.

Methods. Prospective, randomized, controlled trial. We enrolled 117 mechanically ventilated trauma (71) and abdominal (46) surgical patients, older than 18, of both sex. In 57 patients (strict glucose control group) we aimed to maintain the blood glucose level between 4.4 and 6. 1 mmol/L, while in 60 patients (standard glucose control group) it was maintained between 7.8 and 10.0 mmol/L, with the use of continues insulin infusion. Insulin dose adjustments were based on measurements of glucose in capillary blood sample.

Key words: surgical patients; mechanical ventilation; pneumonia; blood glucose; insulin infusion; hospital stay

DETAILED DESCRIPTION:
see brief summary

ELIGIBILITY:
Inclusion Criteria:

* surgical patients
* mechanical ventilated
* both sex
* older than 18

Exclusion Criteria:

* non-surgical patients
* non mechanical ventilated
* younger than 18
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117
Dates: Start 2004-09; Study Completion 2006-07

PRIMARY OUTCOMES:
measurements of glucose in capillary blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Adela Stecher, Principal Investigator — Clinical Centre Ljubljana
Locations (1):
- Clinical Centre Ljubljana, Ljubljana, Ljubljana, Slovenia